CLINICAL TRIAL: NCT00546143
Title: Multi-center, Open-label, Multiple Dose Study in Mild to Moderate Asthmatics (With IgE/Body Weight Combinations Above That in the SmPC Dosing Table) to Determine Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Omalizumab
Brief Title: Safety and Tolerability of Omalizumab in Patients With Mild to Moderate Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025A2208
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Asthma
Keywords: Asthma, anti-immunoglobulin E, omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Omalizumab 900 mg
  Interventions: Drug: Omalizumab
- 2 (Experimental): Omalizumab 1050 mg
  Interventions: Drug: Omalizumab
- 3 (Experimental): Omalizumab 1200 mg
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab
  Other Names: Xolair, IGE025
  Arms: 1
Drug: Omalizumab
  Other Names: Xolair, IGE025
  Arms: 2
Drug: Omalizumab
  Other Names: Xolair, IGE025
  Arms: 3

SUMMARY:
This study will evaluate the safety and efficacy of omalizumab against asthma attacks in mild to moderate allergic asthma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of allergic asthma >= 1 year duration and a history consistent with Step 2 or 3 clinical features from the Global Initiative for Asthma guidelines.
* Eligible baseline serum immunoglobulin E (IgE) levels value and body-weight combinations

Exclusion Criteria:

* Documented medical history of anaphylaxis
* Lung disease other than mild to moderate allergic asthma such as chronic obstructive pulmonary disease (COPD)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of omalizumab assessed by AEs and SAEs

SECONDARY OUTCOMES:
- Pharmacokinetic/pharmacodynamic profile of multiple administrations of omalizumab to patients with mild to moderate allergic asthma - Pre-dose specific IgE levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigative site
Locations (5):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative site, Hamburg
  - Novartis investigative site, Hanover
  - Novartis investigative site, Mainz
- Novartis Investigative site, Bloemfontein, South Africa

REFERENCES:
- [Derived] Kornmann O, Watz H, Fuhr R, Krug N, Erpenbeck VJ, Kaiser G. Omalizumab in patients with allergic (IgE-mediated) asthma and IgE/bodyweight combinations above those in the initially approved dosing table. Pulm Pharmacol Ther. 2014 Aug;28(2):149-53. doi: 10.1016/j.pupt.2014.03.003. Epub 2014 Mar 18. PMID 24657236